CLINICAL TRIAL: NCT02987777
Title: Prognostic Impact of Programmed Death Ligand-1 Expression in Advanced Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2016_0001
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The aim of this study was to assess the frequency of PD-L1 expression in stage III-IV ECs and to investigate its correlation impact with progression-free survival (PFS), and clinicopathological features including microsatellite instability and quantified stromal and intraepithelial tumor-infiltrating CD8+ lymphocytes (TILs)

ELIGIBILITY:
Inclusion Criteria:

* All patients consecutively enrolled from January 2004 to December 2014 treated for Endometrial cancer
* Stage III-IV endometrial cancer with available tissue blocks, including biopsies, hysterectomy specimens and resections of metastatic foci

Exclusion Criteria:

* A patient record captured outside the time frame from January 2004 to December 2014

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records would be extracted from the pathology database of the Lorraine Comprehensive Cancer Center, Nancy, France
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 84 months